CLINICAL TRIAL: NCT04855331
Title: Laparoscopic Versus Open Pancreatoduodenectomy Following Neoadjuvant Chemotherapy for Borderline Resectable Pancreatic Cancer: An Multicenter Open-label Randomized Clinical Trial
Brief Title: Laparoscopic Versus Open Pancreatoduodenectomy Following Neoadjuvant Chemotherapy for BRPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: The Third Affiliated Hospital of Soochow University (Other); Qilu Hospital of Shandong University (Other); West China Hospital (Other); Tongji Hospital (Other); Fujian Provincial Hospital (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, President of Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-5
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Borderline Resectable Pancreatic Cancer
Keywords: Pancreatic Ductal Adenocarcinoma; Neoadjuvant Chemotherapy; Laparoscopic Pancreatoduodenectomy; Safety and Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic pancreatoduodenectomy (Experimental): Laparoscopic pancreatoduodenectomy following neoadjuvant chemotherapy for borderline resectable pancreatic cancer
  Interventions: Procedure: Laparoscopic pancreatoduodenectomy
- Open pancreatoduodenectomy (Active Comparator): Open pancreatoduodenectomy following neoadjuvant chemotherapy for borderline resectable pancreatic cancer
  Interventions: Procedure: Open pancreatoduodenectomy

INTERVENTIONS:
Procedure: Laparoscopic pancreatoduodenectomy — Laparoscopic pancreatoduodenectomy following neoadjuvant chemotherapy for borderline resectable pancreatic cancer.
  Arms: Laparoscopic pancreatoduodenectomy
Procedure: Open pancreatoduodenectomy — Open pancreatoduodenectomy following neoadjuvant chemotherapy for borderline resectable pancreatic cancer.
  Arms: Open pancreatoduodenectomy

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of laparoscopic versus open pancreatoduodenectomy following neoadjuvant chemotherapy for borderline resectable pancreatic cancer

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is one of the most aggressive tumors with an increasing incidence and constitutes the fourth leading cause of cancer-related deaths. Radical resection remains the potential curative treatments for selected patients, and the Miami international evidence-based guidelines suggest that minimally invasive resection is feasible, safe, and oncologically equivalent for PDAC patients compared with open surgery. Furthermore, minimally invasive pancreatomy was associated with better overall and disease-free survival.

However, only 15% to 20% PDAC patients are eligible for upfront surgery at the time of initial diagnosis. For borderline resectable PDAC, studies have confirmed that neoadjuvant therapy can provide more oncological benefits than upfront surgery, such as improved rates of margin-negative resection and decreased incidence of lymph node metastases. Additionally, short-term neoadjuvant therapy has been shown to improve postoperative survival. These findings support the use of short-term neoadjuvant therapy in borderline resectable PDACs, as recommended by the National Comprehensive Cancer Network guidelines.

Neoadjuvant therapy can lead to severe fibrosis in the localized tumor tissue, which may hinder dissection and increase the risk of dangerous and bloody surgery. Furthermore, most anatomically borderline resectable PDACs have a large diameter and are in close proximity to major blood vessels, making the surgical procedure more complex and challenging. To date, there is insufficient evidence to determine the feasibility and safety of minimally invasive pancreatectomy compared to open surgery after neoadjuvant therapy.

This study aims to evaluate the safety and efficacy of laparoscopic pancreatoduodenectomy (LPD) versus open pancreatoduodenectomy (OPD) for borderline resectable PDAC following neoadjuvant chemotherapy (NACT) through a multicenter randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Before neoadjuvant chemotherapy, pancreatic ductal adenocarcinoma was confirmed by pathology;
* According to the guidelines, neoadjuvant chemotherapy should be performed before surgery, including patients with resectable pancreatic cancer (RPC) with high risk factors (biologically borderline resectable), anatomically borderline resectable pancreatic cancer (BRPC) with good physical condition;
* Receive at least 2 cycles of neoadjuvant chemotherapy before radical surgery；
* After neoadjuvant chemotherapy, the patient can be further treated by laparoscopic or open surgery;
* No obvious surgical contraindications, suitable for minimally invasive surgery;
* ECOG score of preoperative physical condition was 0-1;
* No history of preoperative pancreatitis;
* Preoperative PET-CT or other imaging examination did not show distant metastasis;
* The expected postoperative survival time was more than 3 months;
* Be able to comply with research protocol, follow-up plan and other protocol requirements;
* Voluntary participation and signed informed consent.

Exclusion Criteria:

* Neoadjuvant chemotherapy is not suitable before operation according to the guidelines;
* Invasion of adjacent organs, abdominal cavity or distant metastasis was found by introperative exploration;
* Patients requiring total pancreatectomy;
* Severe impairment of heart, liver and kidney function;
* Patients with other malignancies or hematological diseases;
* The patient is pregnant, planning to be pregnant or lactating；
* Before surgery, anti-cancer therapy except neoadjuvant chemotherapy were performed, including interventional chemoembolization, ablation, radiotherapy and molecular targeted therapy;
* Participants in other clinical trials;
* Tumor progression occurred during neoadjuvant chemotherapy. After neoadjuvant chemotherapy, patients failed reach the standard of laparoscopic surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 90 days after the surgery
  The specific postoperative complications of pancreatic surgery include postoperative pancreatic fistula, postoperative hemorrhage and gastroparesis. Other common postoperative complications include abdominal infection, incision nonunion and so on. The degree of complications was evaluated by Clavien-Dindo grading system.

SECONDARY OUTCOMES:
Length of stay | 90 days after the surgery
  The length of hospital stay from the end of surgery to discharge or death. The length of hospital stay for readmission after discharge is not included.
Operation time | 1 day
  The time from the beginning to the end of the surgery.
R0 resection rate | 30 days after the surgery
  Postoperative pathology confirmed that there were no tumor cells in the tissue within 1 mm from the surgical margin.
The 90 days readmission rate | 90 days after the surgery
  The rate of rehospitalization within 90 days after surgery due to aggravation.
The 90 days mortality rate after operation | 90 days after the surgery
  The mortality within 90 days after surgery.

OTHER OUTCOMES:
Recurrence free survival | up to 5 years after the surgery
  The time from surgery until tumor recurrence, death or the last follow-up time.
Overall survival | up to 5 years after the surgery
  The time from surgery until death or the last follow-up time.
Postoperative quality of life | up to 5 years after the surgery
  Postoperative quality of life was assessed by the European Organization for Research and Treatment of Cancer (EORTC) quality of life scale QLQ-C30 and pancreatic cancer quality of life specific scale QLQ-PAN26.

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, MD, PhD, Principal Investigator — Fudan University; Xiaowu Xu, MD, Study Director — Fudan University
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mokdad AA, Minter RM, Zhu H, Augustine MM, Porembka MR, Wang SC, Yopp AC, Mansour JC, Choti MA, Polanco PM. Neoadjuvant Therapy Followed by Resection Versus Upfront Resection for Resectable Pancreatic Cancer: A Propensity Score Matched Analysis. J Clin Oncol. 2017 Feb 10;35(5):515-522. doi: 10.1200/JCO.2016.68.5081. Epub 2016 Sep 30. PMID 27621388
- [Background] Sugimoto M, Takahashi N, Farnell MB, Smyrk TC, Truty MJ, Nagorney DM, Smoot RL, Chari ST, Carter RE, Kendrick ML. Survival benefit of neoadjuvant therapy in patients with non-metastatic pancreatic ductal adenocarcinoma: A propensity matching and intention-to-treat analysis. J Surg Oncol. 2019 Nov;120(6):976-984. doi: 10.1002/jso.25681. Epub 2019 Aug 26. PMID 31452208
- [Background] Versteijne E, Suker M, Groothuis K, Akkermans-Vogelaar JM, Besselink MG, Bonsing BA, Buijsen J, Busch OR, Creemers GM, van Dam RM, Eskens FALM, Festen S, de Groot JWB, Groot Koerkamp B, de Hingh IH, Homs MYV, van Hooft JE, Kerver ED, Luelmo SAC, Neelis KJ, Nuyttens J, Paardekooper GMRM, Patijn GA, van der Sangen MJC, de Vos-Geelen J, Wilmink JW, Zwinderman AH, Punt CJ, van Eijck CH, van Tienhoven G; Dutch Pancreatic Cancer Group. Preoperative Chemoradiotherapy Versus Immediate Surgery for Resectable and Borderline Resectable Pancreatic Cancer: Results of the Dutch Randomized Phase III PREOPANC Trial. J Clin Oncol. 2020 Jun 1;38(16):1763-1773. doi: 10.1200/JCO.19.02274. Epub 2020 Feb 27. PMID 32105518
- [Background] Reni M, Balzano G, Zanon S, Zerbi A, Rimassa L, Castoldi R, Pinelli D, Mosconi S, Doglioni C, Chiaravalli M, Pircher C, Arcidiacono PG, Torri V, Maggiora P, Ceraulo D, Falconi M, Gianni L. Safety and efficacy of preoperative or postoperative chemotherapy for resectable pancreatic adenocarcinoma (PACT-15): a randomised, open-label, phase 2-3 trial. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):413-423. doi: 10.1016/S2468-1253(18)30081-5. Epub 2018 Apr 4. PMID 29625841
- [Background] Jang JY, Han Y, Lee H, Kim SW, Kwon W, Lee KH, Oh DY, Chie EK, Lee JM, Heo JS, Park JO, Lim DH, Kim SH, Park SJ, Lee WJ, Koh YH, Park JS, Yoon DS, Lee IJ, Choi SH. Oncological Benefits of Neoadjuvant Chemoradiation With Gemcitabine Versus Upfront Surgery in Patients With Borderline Resectable Pancreatic Cancer: A Prospective, Randomized, Open-label, Multicenter Phase 2/3 Trial. Ann Surg. 2018 Aug;268(2):215-222. doi: 10.1097/SLA.0000000000002705. PMID 29462005
- [Background] Philip PA, Lacy J, Portales F, Sobrero A, Pazo-Cid R, Manzano Mozo JL, Kim EJ, Dowden S, Zakari A, Borg C, Terrebonne E, Rivera F, Sastre J, Bathini V, Lopez-Trabada D, Asselah J, Saif MW, Shiansong Li J, Ong TJ, Nydam T, Hammel P. Nab-paclitaxel plus gemcitabine in patients with locally advanced pancreatic cancer (LAPACT): a multicentre, open-label phase 2 study. Lancet Gastroenterol Hepatol. 2020 Mar;5(3):285-294. doi: 10.1016/S2468-1253(19)30327-9. Epub 2020 Jan 14. PMID 31953079
- [Background] de Rooij T, van Hilst J, van Santvoort H, Boerma D, van den Boezem P, Daams F, van Dam R, Dejong C, van Duyn E, Dijkgraaf M, van Eijck C, Festen S, Gerhards M, Groot Koerkamp B, de Hingh I, Kazemier G, Klaase J, de Kleine R, van Laarhoven C, Luyer M, Patijn G, Steenvoorde P, Suker M, Abu Hilal M, Busch O, Besselink M; Dutch Pancreatic Cancer Group. Minimally Invasive Versus Open Distal Pancreatectomy (LEOPARD): A Multicenter Patient-blinded Randomized Controlled Trial. Ann Surg. 2019 Jan;269(1):2-9. doi: 10.1097/SLA.0000000000002979. PMID 30080726
- [Background] Croome KP, Farnell MB, Que FG, Reid-Lombardo KM, Truty MJ, Nagorney DM, Kendrick ML. Total laparoscopic pancreaticoduodenectomy for pancreatic ductal adenocarcinoma: oncologic advantages over open approaches? Ann Surg. 2014 Oct;260(4):633-8; discussion 638-40. doi: 10.1097/SLA.0000000000000937. PMID 25203880
- [Background] Wang M, Li D, Chen R, Huang X, Li J, Liu Y, Liu J, Cheng W, Chen X, Zhao W, Li J, Tan Z, Huang H, Li D, Zhu F, Qin T, Ma J, Yu G, Zhou B, Zheng S, Tang Y, Han W, Meng L, Ke J, Feng F, Chen B, Yin X, Chen W, Ma H, Xu J, Liu Y, Lin R, Dong Y, Yu Y, Liu J, Zhang H, Qin R; Minimally Invasive Treatment Group in the Pancreatic Disease Branch of China's International Exchange and Promotion Association for Medicine and Healthcare (MITG-P-CPAM). Laparoscopic versus open pancreatoduodenectomy for pancreatic or periampullary tumours: a multicentre, open-label, randomised controlled trial. Lancet Gastroenterol Hepatol. 2021 Jun;6(6):438-447. doi: 10.1016/S2468-1253(21)00054-6. Epub 2021 Apr 27. PMID 33915091
- [Background] Asbun HJ, Moekotte AL, Vissers FL, Kunzler F, Cipriani F, Alseidi A, D'Angelica MI, Balduzzi A, Bassi C, Bjornsson B, Boggi U, Callery MP, Del Chiaro M, Coimbra FJ, Conrad C, Cook A, Coppola A, Dervenis C, Dokmak S, Edil BH, Edwin B, Giulianotti PC, Han HS, Hansen PD, van der Heijde N, van Hilst J, Hester CA, Hogg ME, Jarufe N, Jeyarajah DR, Keck T, Kim SC, Khatkov IE, Kokudo N, Kooby DA, Korrel M, de Leon FJ, Lluis N, Lof S, Machado MA, Demartines N, Martinie JB, Merchant NB, Molenaar IQ, Moravek C, Mou YP, Nakamura M, Nealon WH, Palanivelu C, Pessaux P, Pitt HA, Polanco PM, Primrose JN, Rawashdeh A, Sanford DE, Senthilnathan P, Shrikhande SV, Stauffer JA, Takaori K, Talamonti MS, Tang CN, Vollmer CM, Wakabayashi G, Walsh RM, Wang SE, Zinner MJ, Wolfgang CL, Zureikat AH, Zwart MJ, Conlon KC, Kendrick ML, Zeh HJ, Hilal MA, Besselink MG; International Study Group on Minimally Invasive Pancreas Surgery (I-MIPS). The Miami International Evidence-based Guidelines on Minimally Invasive Pancreas Resection. Ann Surg. 2020 Jan;271(1):1-14. doi: 10.1097/SLA.0000000000003590. PMID 31567509
- [Background] Chawla A, Molina G, Pak LM, Rosenthal M, Mancias JD, Clancy TE, Wolpin BM, Wang J. Neoadjuvant Therapy is Associated with Improved Survival in Borderline-Resectable Pancreatic Cancer. Ann Surg Oncol. 2020 Apr;27(4):1191-1200. doi: 10.1245/s10434-019-08087-z. Epub 2019 Dec 4. PMID 31802297
- [Background] Roland CL, Yang AD, Katz MH, Chatterjee D, Wang H, Lin H, Vauthey JN, Pisters PW, Varadhachary GR, Wolff RA, Crane CH, Lee JE, Fleming JB. Neoadjuvant therapy is associated with a reduced lymph node ratio in patients with potentially resectable pancreatic cancer. Ann Surg Oncol. 2015 Apr;22(4):1168-75. doi: 10.1245/s10434-014-4192-6. Epub 2014 Oct 29. PMID 25352267
- [Background] Miyasaka Y, Ohtsuka T, Kimura R, Matsuda R, Mori Y, Nakata K, Kakihara D, Fujimori N, Ohno T, Oda Y, Nakamura M. Neoadjuvant Chemotherapy with Gemcitabine Plus Nab-Paclitaxel for Borderline Resectable Pancreatic Cancer Potentially Improves Survival and Facilitates Surgery. Ann Surg Oncol. 2019 May;26(5):1528-1534. doi: 10.1245/s10434-019-07309-8. Epub 2019 Mar 13. PMID 30868514